CLINICAL TRIAL: NCT04261556
Title: Innovative Protocol Targeting Cognitive Dysfunction in Multiple Sclerosis: tDCS to Enhance Cognitive Training in a Randomized, Double-blind, Controlled, Exploratory Pilot Study
Brief Title: tDCS to Enhance Cognitive Training in Multiple Sclerosis
Acronym: REHACOG-MS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to organizing difficulties after COVID-19 pandemic
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REHACOG-MS
Record Dates: First submitted 2019-12-04; First posted 2020-02-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Relapsing remitting multiple sclerosis; Cognitive training; Cognitive rehabilitation; Cognitive remediation; Neuromodulation; Transcranial direct current stimulation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS + CCT (Experimental): 40 min/day of computerised cognitive training (CCT) + 20 min/day of real anodal transcranial direct current stimulation (tDCS).
  In the first 20 min of the 40 min-intervention, tDCS and CCT will be provided simultaneously.
  Interventions: Device: Real tDCS + CCT
- Sham tDCS + CCT (Sham Comparator): 40 min/day of CCT + 20 min/day of apparent (sham) tDCS. In the first 20 min of the 40 min-intervention, tDCS and CCT will be provided simultaneously.
  Interventions: Device: Sham tDCS + CCT

INTERVENTIONS:
Device: Real tDCS + CCT — 40 min/day of computerised cognitive training (CCT) + 20 min/day of real anodal transcranial direct current stimulation (tDCS).
  In the first 20 min of the 40 min-intervention, real anodal tDCS and CCT will be provided simultaneously.
  Arms: Real tDCS + CCT
Device: Sham tDCS + CCT — 40 min/day of computerised cognitive training (CCT) + 20 min/day of apparent (sham) tDCS.
  In the first 20 min of the 40 min-intervention, sham tDCS and CCT will be provided simultaneously.
  Arms: Sham tDCS + CCT

SUMMARY:
Expected results: an improvement in cognitive performance in both groups, boosted in the experimental arm and not confined to general frontal-cognitive abilities; potential changes would be reflected also by neurophysiological measures and in QoL.

Discussion: Investigators hope to provide additional treatment tools for RRMS subjects, with a medium-long term efficacy and an extensive effect. This exploratory pilot study will help to set the rationale for future studies, providing preliminary data useful for selecting the best primary outcome and for calculating a better sample size.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically definite diagnosis of relapsing remitting MS (RRMS);
* Male or female subjects, 18 to 65 years old;
* Expanded Disability Status Scale (EDSS) score ranging from 0 to 5.5 (included);
* Predominant deficits in either attention/information processing;
* Fluent Italian speakers;
* Normal or corrected-to-normal vision;
* Ability to understand the purpose and risk of the study and provide signed informed consent.

Exclusion Criteria:

* MS patients in different phase of the disease (as primary/secondary progressive MS; benign MS) or Clinical Isolated Syndrome (CIS) patients;
* Exclusive cognitive impairment in different domains (e.g., memory);
* CT/neuromodulation program ongoing or in the preceding 6 months;
* Clinical exacerbations, neuroradiological activity of the disease, modification of EDSS score and disease modifying treatments/steroids during the last 3 months preceding study enrolment;
* Significant medical disorders or other major systemic, psychiatric, neurological disorders or alcohol/substance abuse that could interfere with cognitive functioning;
* Antidepressant/psychoactive drugs in the past 3 months;
* Contraindications to tDCS (intracranial metallic plates, implanted devices, skin disease, superficial injury and fracture or infraction of skull in the stimulation area, epilepsy, pregnancy, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Symbol Digit Modalities Test (SDMT) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Change in target cognitive test assessing information processing (i.e., SDMT)
Change in Paced Auditory Serial Addition Test (PASAT) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Change in target cognitive test assessing information processing (i.e., PASAT)
Change in Wisconsin Card Sorting Test (WCST) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Change in target cognitive test assessing frontal executive functions (i.e., WCST)
Change in Stroop test | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Change in target cognitive test assessing frontal executive functions (i.e., Stroop test)
Change in Digit Spans | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Change in target cognitive tests assessing information processing and frontal executive functions (i.e., digit spans)

SECONDARY OUTCOMES:
Number of sessions done by esch participants (Feasibility) | Day 0 (baseline, T0), Week 2 (end of treatment, T1)
  Overall compliance of the protocol, assessed by number of sessions done by esch participants (Feasibility)
Number tDCS-related of discomfort or side effects experienced by each participants (Safety) | Day 0 (baseline, T0), Week 2 (end of treatment, T1)
  Any tDCS-related discomfort or side effect after each daily session
Changes in Brief Repeatable Battery of Neuropsychological Tests (BRBN-T) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Changes in single subtest of the BRBN-T
Changes in Beck Depression Inventory (BDI) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  21-question multiple-choice self-report inventory, higher score means worse depressive score.
Changes in Expanded Disability Status Scale (EDSS) measurements | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  10 points scale, higher score means worse disease progression.
Changes in Multiple Sclerosis Functional Composite (MFSC) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Three component parts, higher scores means worse functional symptoms.
Changes in Modified Fatigue Impact Scale (MFIS) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. higher scores indicate a greater impact of fatigue
Changes in Multiple Sclerosis Quality of Life (MSQOL-54) | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores.
Changes in alpha oscillations measured with Electroencephalogram (EEG) Resting State From Baseline | Day 0 (baseline, T0), Week 2 (end of treatment, T1), Follow-up at 3 months (FU3) and follow-up at 6 months (FU6)
  Comparison of alpha oscillation power from resting state EEG recordings on the first and last day of protocol. EEG data also recorded at 3- and 6-month follow up visits. Each of the four EEG recordings will serve to analyze alpha frequency activity for derivation of EEG biomarkers in this observational pilot study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano-Bicocca, Monza, Italy

IPD SHARING:
Plan to Share IPD: No